CLINICAL TRIAL: NCT06982417
Title: InsightRP2: a Global Patient Registry for RP2-associated Retinitis Pigmentosa
Brief Title: InsightRP2 Registry
Status: Recruiting | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Nina Bogershausen, MD, University of Göttingen
Other Study IDs: 11/11/24
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: RP2-associated Retinitis Pigmentosa; X-Linked Retinitis Pigmentosa (XLRP); Retinitis Pigmentosa 2
Keywords: RP2, Retinitis pigmentosa, RP2-associated Retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa 2; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Retinitis pigmentosa due to a variant / mutation in the RP2 gene: A molecular genetic diagnosis involving a heterozygous or hemizygous variant in RP2 and a written informed consent to participate are required for access to the registry questionnaire. Patients of all ages meeting the above criteria will be allowed to participate.

SUMMARY:
InsightRP2 is a secure online patient registry specific to RP2-associated retinitis pigmentosa (RP). It is our goal to further the scientific understanding of this rare disease and to support research in to a gene therapy for RP2-associated RP.

We collect medical, genetic and imaging data from people affected by RP2-associated RP and will coduct a natural history study as well as image analysis studies.

DETAILED DESCRIPTION:
There is currently no specific patient registry for RP2-associated retinitis pigmentosa. Due to the rarity of the disease, only a few patients with this disease are seen at various care sites, making clinical care and diagnosis very challenging. In addition, there are numerous knowledge gaps regarding the course of the disease, the disease mechanisms and therapeutic approaches, which poses additional challenges for patient care. Understanding and future treatment of RP2-associated RP is crucial due to its early onset and rapid progression. There is an urgent need for targeted research to develop effective therapies.

At the Institute of Human Genetics Göttingen, we have set ourselves the goal of investigating the disease mechanisms of RP2-associated RP and contributing to the long-term development of a therapy for this rare disease.

For this purpose, we have set up a patient registry specifically for RP2-associated RP. The registry is fully online, using a secure REDCap-based database hosted at the University Medical Center Göttingen. The medical data collected will enable us to conduct studies on the natural history, mutation distribution and possible genotype-phenotype correlations of this disease. In addition, the collection of medical image data will enable evaluation for the purpose of improving diagnostic processes and supporting therapeutic studies. Last but not least, we aim to form a patient collective who can be offered participation in possible therapy studies at a later date.

We will collect retrospective data, however patient's might be recontacted at a later timepoint, which is why we have designated the time perspective as "other" in the description of the study design.

ELIGIBILITY:
Inclusion Criteria:

* A molecular genetic diagnosis involving a heterozygous or hemizygous variant in RP2 and a written informed consent to participate are required for access to the registry questionnaire. Patients of all ages meeting the above criteria will be allowed to participate. As documentation will be in English and German, those who can navigate these pages will be included.

Exclusion Criteria:

* Patients with evidence of non-RP2 molecular genetic diagnoses will be excluded. Collection of data and further analysis will not be possible without the consent of the patient or legal guardian. Patients who cannot navigate registry documentation in English or German will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals affected by RP2-associated Retinitis pigmentosa worldwide.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2045-05-01 (Estimated); Study Completion 2045-05-01 (Estimated)

PRIMARY OUTCOMES:
Genotype-phenotype correlation age of onset | 1 year
  Influence of variant type on age of onset
Phenotype-genotype correlation progression | 20 years
  Influence of variant type on disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will be collected over a longer period of time. IPD will be shared as a supplementary information to a publication and made accessible in an open access journal. Informed consent information is freely available in the registry or via our homepage (see links).

REFERENCES:
- See also: Homepage containing information about the InsightRP2 study and registry, as well as links to access the informed consent depending on the participant's age. — https://www.humangenetik-umg.de/en/research/wollnik-research-group/insightrp2/

DOCUMENTS (1):
  • Study Protocol (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT06982417/Prot_000.pdf